CLINICAL TRIAL: NCT05294900
Title: Phase II Trial of Neoadjuvant Therapy With Paclitaxel and Carboplatin in Operable Locally Advanced Head and Neck Cancer Patients (NEOS)
Brief Title: Trial of Neoadjuvant Therapy With Paclitaxel and Carboplatin in Operable Locally Advanced Head and Neck Cancer Patients
Acronym: NEOS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-3771-003
Record Dates: First submitted 2022-03-15; First posted 2022-03-24 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: HNSCC; Neo-adjuvant chemotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — CP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- paclitaxel/carboplatin (Experimental): paclitaxel+carboplatin
  Interventions: Drug: paclitaxel/carboplatin

INTERVENTIONS:
Drug: paclitaxel/carboplatin — Induction chemotherapy : total 2 cycle every 3weeks as below:
  * Paclitaxel 175mg/m2
  * Carboplatin AUC5

SUMMARY:
- Objective: Primary objective: To evaluate the major pathologic response (mPR) of locally advanced head and neck cancer after paclitaxel and carboplatin-induction chemotherapy followed by surgery.

Secondary objective: To evaluate the efficacy and safety of induction chemotherapy. Outcome metrics: Local relapse rate (LRR), Relapse-free survival (RFS), Overall survival (OS), Adverse reactions according to CTCAE 5.0 Exploratory Purpose: To evaluate changes in circulating tumor cells (CTC) and immunodynamics before and after paclitaxel and carboplatin-induction chemotherapy through blood, biopsy specimens, and surgical specimen analysis.

* background :

  * Chemoradiation (CRT) or chemotherapy (Induction Chemotherapy (IC) + CRT) after induction chemotherapy has been performed for locally advanced head and neck cancer that cannot be operated immediately or for organ function preservation. .
  * The efficacy of induction chemotherapy before chemotherapy has been controversial because the results of several phase 3 clinical studies are inconsistent. At present, it is difficult to assert the superiority of either the addition of induction chemotherapy or radiation therapy alone, but in certain subgroups (advanced N stage such as N2c/N3) induction chemotherapy is a useful option to lower distant metastases. I can do it.
  * As a result of the TAX324 clinical trial, when weekly carboplatin-based chemotherapy or surgery was performed after adjuvant Docetaxel + Cisplatin + 5FU chemotherapy, overall survival was improved compared to Cisplatin + 5FU (HR 0.7, p=0.0058), It resulted in improvement of institutional retention rate (3 year LFS: 52% vs 32%). However, it is difficult to apply this TPF therapy to all patients in actual clinical practice due to the toxicity (neutropenia, nephrotoxicity) and the limitation of anticancer radiation.
  * In a retrospective study, in the case of adjuvant paclitaxel + carboplatin, there was no difference in progression-free survival compared to TPF (p=0.15), and there was no statistically significant decrease in the local recurrence rate (HR 0.27, p = 0.04). Confirmed.
  * Therefore, in this study, when paclitaxel and carboplatin-induction chemotherapy followed by surgery and chemotherapy after surgery, compared to standard TPF-induced chemotherapy, it is expected that the clinical outcome will be improved with less toxicity.
* Hypothesis: Paclitaxel and carboplatin-induction chemotherapy followed by surgery, followed by chemo-radiation after surgery according to standard guidelines Compared with the existing standard treatment (TCF), improvement of clinical outcome with less toxicity
* Study procedure

  * Induction chemotherapy Paclitaxel 175mg/m2 + Carboplatin AUC5 (calculated by Cockcroft - Gault formula) Combination therapy A total of 2 intravenous infusions every 3 weeks Surgery performed within 2-9 weeks after induction chemotherapy
  * surgery The surgery in this study means a complete resection for the purpose of a complete cure, and aims for a minimally invasive surgery.

DETAILED DESCRIPTION:
o Induction chemotherapy Paclitaxel 175mg/m2 + Carboplatin AUC5 (calculated by Cockcroft - Gault formula) Combination therapy A total of 2 intravenous infusions every 3 weeks"

ELIGIBILITY:
Inclusion

1. A patient whose potentially surgical, teletransfer-free HNSCC of oral, hypodermic, occipital, and larynx has been tissue-confirmed Oral cancer of III-IV, laryngeal cancer, hypodermic cancer, HPV-negative head cancer II-III HPV positive head cancer
2. A disease that can be measured, defined as a lesion that can be accurately measured pursuant to RECIST 1.1
3. Where the candidate subject to the test prepares the consent of the person subject to the test after obtaining approval required by region before the commencement of any plan-related procedures, including screening evaluation
4. Adult men and women over 20 years old at the time of participation in clinical trials
5. Eastern Cancer Cooperation Research Group (Eastern Cooperative Oncology Group, ECOG) Activity Status 0 or 1
6. A patient with a life expectancy of at least 12 weeks
7. Proper and normal organ and bone marrow functions as defined below:

   * hemoglobin test 9.0 g/dL
   * Absolute neutropenic number (ANC) set 109/L (1500 per mm3)
   * Platelet count 75,000 per mm3
   * 1.5 times the total ULN of serum biliubine test institution
   * 2.5 times the ULN of the AST (SGOT)/ALT (SGPT) test institute.
   * Creatinine cleaning rate measured by 24-hour urine collection samples > 40 mL/min or calculated by Cockcroft Gault formula (Cockcroft and Gault 1976) >40 mL/min:
8. Women who have evidence after menopause or pre-menopausal women whose urine or serum pregnancy test results are negative. Women who have amenorrhea for 12 months without other medical reasons are considered after menopause. The following age requirements apply:

   * Even under the age of 50, she is in amenorrhea for at least 12 months after discontinuing exogenous hormone treatment, and if the LH and FSH levels are the menopause levels of the test institute, or if she underwent a surgical infertility operation (bilateral ovarian resection or complete hysterectomy), she is considered a menopause woman.
   * Women who have been in amenorrhea for at least 12 months after stopping all external hormone treatment, or whose last menstrual period is at least a year before and after radiation-induced menopause, or more than a year after chemotherapy induced menopause or who have undergone surgical infertility (bilateral ovarian resection, bilateral tubulectomy, or full hysterectomy) are considered women with menopause.

Exclusion

1. Direct involvement in the planning and/or implementation of this clinical trial
2. Patients with nasopharyngeal cancer
3. A patient who has experienced previous treatment for head and neck cancer (including a history of radiation treatment)
4. Patients who have participated in other clinical trials using clinical drugs within the past month
5. A patient registered simultaneously in a clinical trial other than an observation (non-mediate) clinical trial or an intermediary clinical trial tracer
6. Patients who need to use additional chemotherapy, clinical medicine, biological medicine, or hormone therapy for chemotherapy: Provided, That the simultaneous use of hormone therapy (e.g. hormone replacement therapy) for conditions unrelated to cancer is allowed.
7. The toxicity of at least NCI CTCAE Level 2 of the previous anti-cancer treatment, which has not yet been resolved: Provided, That laboratory values defined as hair loss, vitiligo, and selection criteria shall be excluded.
8. Neuropathy of grade 2 or higher is determined after consultation with a clinical trial doctor on a case-by-case basis.
9. Patients with irreversible toxicity that is not expected to worsen due to the administration of clinical trials can participate in the test only after consultation with a clinical trial doctor.
10. Patients who undergo a major operation (according to the tester's definition) within 28 days before the initial administration of clinical medication. Note: Local surgery on independent lesions for the purpose of conventional treatment is acceptable.
11. Intractable diseases, but not limited to the following: ongoing or active infections; symptom congestive heart failure; uncontrolled high blood pressure; unstable angina; heart veins; epileptic lung disease; Major chronic gastrointestinal conditions with diarrhea; All mental/social conditions that may restrict compliance with clinical trial requirements or significantly increase the risk of adverse reactions or hinder the subject's ability to write consent
12. A patient who has a history of another primary malignant tumor: Provided, That the following shall not apply:

    * A past malignant tumor that was treated for the purpose of complete cure and has no history of a known active disease within five years before the initial administration of clinical medication and has a low risk of recurrence
    * non-black skin cancer treated properly or malignant black spots without evidence of disease
    * Carcinoma that has been properly treated and has no evidence of disease
13. History of active primary immune deficiency
14. Women who are currently pregnant or breastfeeding or fertile men and women who are not willing to use effective contraception from the time of screening to 180 days after the end of clinical treatment
15. Patients who are known to be allergic or irritable to clinical trials drugs or their siblings
16. Patients who are not suitable to participate in clinical trials and are not expected to comply with clinical trial procedures, restrictions, and requirements according to the judgment of the tester

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response(mPR) | up to 9weeks after completion of the induction chemotherapy

SECONDARY OUTCOMES:
Loco-regional relapse rate(LRR) | up to 9weeks after completion of the induction chemotherapy
Relapse-free survival(RFS) | Up to 1 years
Overall survival (OS) | Up to 1 years

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No